CLINICAL TRIAL: NCT06084728
Title: 3D Ultrasound and Color Doppler Studies of the Clitoris in Pregnant Women
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Other Study IDs: 72
Record Dates: First submitted 2023-10-01; First posted 2023-10-16 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Clitoris Vascularity
MeSH Terms: interventions — Ultrasonography, Doppler, Color; Echocardiography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women: 30 pregnant women.
  Interventions: Diagnostic Test: Color Doppler ultrasonography
- Non-pregnant women: 30 non pregnant women as control group
  Interventions: Diagnostic Test: Color Doppler ultrasonography

INTERVENTIONS:
Diagnostic Test: Color Doppler ultrasonography — in a longitudinal plane, the dorsal clitoral artery, which is sampled on the outer surface of the clitoral body as previously described. With the same longitudinal approach, the terminal branch of the posterior labial artery (a branch of the internal pudendal artery) was visualized posterolaterally to the labia majora
  Other Names: Doppler

SUMMARY:
Patients will be divided into two groups:

Group A: 30 pregnant women Group B: 30 non pregnant women as control group.

All patients will be subjected to the following:

1. Interview with women for detailed history taking and explaining the research. A written Consent will be obtained from them before their enrollment into the study.
2. To ensure standard conditions, the subjects will lie in a recumbent position and were evaluated between 08.00 and 11.00 a.m. To avoid anyexternal genital stimulation, subjects will be asked not to wear trousers or cross their legs on the morning of the ultrasound examination.
3. Furthermore, in order to minimize external effects on blood flow, all women will be scanned in a noiseless room with constant heat and light

DETAILED DESCRIPTION:
Patients will be divided into two groups:

Group A: 30 pregnant women Group B: 30 non pregnant women as control group. Translabial ultrasound scanning will be performed for each woman with Sonographic measurements of the clitoral volume and labia minora thickness performed by using a RSP-16 multi frequency transducer. The transducer will be placed on the upper part of the vulva to assess the clitoris in a transverse section and on the labia majora for the sagittal view. To prevent artifacts, care will be taken to avoid excessive pressure on the clitoris. The clitoris was studied where the paired corpora join in a single body that projects into the glans. Volumes were measured by reporting length, width, and depth assuming the form to be an ellipsoid: V = π/6 × D1 × D2 × D3, where D1, D2, and D3 are the maximal longitudinal, anteroposterior, and transverse diameter, respectively. The same transducer will be sagittally placed on each labium major to measure labia minora thickness, ensuring that the minimum possible pressure is applied with the ultrasound probe on the skin.

Color Doppler ultrasonography will be used to identify, in a longitudinal plane, the dorsal clitoral artery, which is sampled on the outer surface of the clitoral body as previously described. With the same longitudinal approach, the terminal branch of the posterior labial artery (a branch of the internal pudendal artery) will be visualized posterolaterally to the labia majora (at about 2 cm from the clitoral hood).

ELIGIBILITY:
Inclusion Criteria:

* Both pregnant and non pregnant women between 18 and 45 years old

Exclusion Criteria:

* Women with genital anomalies
* Virgins
* Women with gynecological disorders as endometriosis or pelvic pathology causing pelvic congestion
* Genital inflammations or mases Neurological or vascular disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Both pregnant and non pregnant women between 18 and 45 years old
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The peak systolic velocity of the clitoreal artery | At time of Doppler assessment
  The peak systolic velocity of the clitoreal artery using Doppler machine to measure Blood supply to the body of clitoris in cm/second
The pulsatility index of clitoreal artery | At time of Doppler assessment
  The pulsatility index of clitoreal artery using Doppler machine to measure Blood supply to the body of clitoris in cm/second

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Seleem, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No